CLINICAL TRIAL: NCT00718471
Title: Acute STEMI Treated With Primary Angioplasty and Intravenous 0.5 mg/kg Lovenox or UFH to Lower Ischemic and Bleeding Events
Brief Title: STEMI Treated With Primary Angioplasty and Intravenous Lovenox or Unfractionated Heparin (UFH)
Acronym: ATOLL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P071101; EUDRACT: 2007-007676-42
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Primary PCI - STEMI
Keywords: STEMI; Primary PCI; Anticoagulation
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Enoxaparin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Enoxaparin
  Interventions: Drug: Enoxaparin
- 2 (Active Comparator): UFH
  Interventions: Drug: UFH (unfractionated heparin)

INTERVENTIONS:
Drug: Enoxaparin — ENOXAPARIN IV 0.5 mg.kg
  Arms: 1
Drug: UFH (unfractionated heparin) — UFH IV 50-70 IU if GP IIbIIIa or 70-100IU if no GP IIbIIIa
  Arms: 2

SUMMARY:
Randomized evaluation of enoxaparin (0.5mg/kg IV) versus UFH (50-70IU/kg with GPIIb/IIIa inhibitors; 70-100IU without GPIIb/IIIa inhibitors). Anticoagulation can be continued after the procedure using the same agents as those allocated per randomization (enoxaparin SC, UHF IV or SC)

DETAILED DESCRIPTION:
This study is a prospective, multicenter, multinational, randomized, active-control arm trial. The study population consists of subjects with ST-segment elevation MI who are randomized within 24 hours of symptom onset. Subjects presenting between 12 and 24 hours of symptom onset should present with recurrent or persisting chest pain and/or recurrent or persisting ST elevation suggesting ongoing ischemia, and an indication of primary PCI.

Approximately 850 subjects will be enrolled at approximately 50 sites in several countries including Austria, France, Germany and the United States. Informed consent will be obtained from subjects meeting all inclusion and no exclusion criteria prior to any study related procedures. Subjects will be randomized and begin treatment in the Emergency Department or in the ambulance or in the hospital room if in-patient. Eligible subjects will be randomized (1:1) to receive either UFH IV bolus (ACT-adjusted) or enoxaparin 0.50 mg/kg IV bolus without monitoring. Randomization to treatment group will be performed using an interactive voice response system (IVRS). All treatment groups will be given aspirin (160 to 500 mg/day according to local practice) and clopidogrel (300 to 900mg as loading dose according to local practice). All other concomitant medications will be consistent with local standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age.
2. Has experienced continuous ischemic (cardiac) symptoms for at least 20 minutes.
3. Has onset of symptoms of qualifying acute MI within the past 24 hours, and planned for primary PCI. Patients presenting between 12 and 24 hours of symptom onset should still have an indication for primary PCI, i.e. persistent ischemic symptom and/or persistent or recurrent ST elevation
4. Has an ECG indicative of an acute STEMI showing:

   * ≥ 2 mm ST elevation in 2 or more contiguous precordial ECG leads (anterior infarction); or
   * ≥ 1 mm ST elevation in 2 or more contiguous limb ECG leads (other infarction); or
   * New or presumably new left bundle branch block (LBBB)
5. Shock patients are eligible (but not patients with prolonged cardiac arrest)
6. Be willing to provide informed consent (informed consent may be provided by a legally authorized representative if the patient is not able to provide it).
7. Agree to comply with all protocol-specified procedures, including protocol-mandated follow-up

Exclusion Criteria:

1. Use of UFH or LMWH or any other anticoagulant agent (Vit K antagonists, fondaparinux, bivalirudin) within 48 hours prior to randomization
2. Thrombolytic therapy within the previous 48 hours
3. Known or suspected pregnancy in women of childbearing potential
4. History of hypersensitivity or contraindication to heparin or LMWH
5. Contraindication to primary PCI or any excessive bleeding risk (e.g. recent surgery) or suspected active internal bleeding
6. Coexistent condition associated with a limited life expectancy at short term (e.g. advanced cancer)
7. Prolonged (> 10 minutes) cardiopulmonary resuscitation (CPR)
8. Treatment with other investigational agents or devices within the previous 30 days, planned use of investigational drugs or devices, or previous enrolment in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 910 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
All-cause mortality or Complications of MI or Procedure failure or Non-CABG major bleeding during hospitalization | administration

SECONDARY OUTCOMES:
major bleeding during hospitalization | during hospitalization and at 6 months
the ischemic end-point of death, reinfarction, refractory ischemia and/or urgent revascularization | day30 and 6 months
efficacy objectives are each individual ischemic endpoint of the primary objective as well as the composite ischemic end-point of death, complications of MI or procedure failure. | day 30 and 6 months
the composite of major and minor bleeding during hospitalization | during hospitalization and months 6

CONTACTS AND LOCATIONS:
Overall Officials: Gilles MONTALESCOT, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- La Pitié-Salpétrière Hospital - Cardiology department, Paris, France

REFERENCES:
- [Result] Montalescot G, Zeymer U, Silvain J, Boulanger B, Cohen M, Goldstein P, Ecollan P, Combes X, Huber K, Pollack C Jr, Benezet JF, Stibbe O, Filippi E, Teiger E, Cayla G, Elhadad S, Adnet F, Chouihed T, Gallula S, Greffet A, Aout M, Collet JP, Vicaut E; ATOLL Investigators. Intravenous enoxaparin or unfractionated heparin in primary percutaneous coronary intervention for ST-elevation myocardial infarction: the international randomised open-label ATOLL trial. Lancet. 2011 Aug 20;378(9792):693-703. doi: 10.1016/S0140-6736(11)60876-3. PMID 21856483
- [Derived] Silvain J, O'Connor SA, Yan Y, Kerneis M, Hauguel-Moreau M, Zeitouni M, Overtchouk P, Ankri A, Brugier D, Vicaut E, Ecollan P, Galier S, Collet JP, Montalescot G; ATOLL Investigators. Biomarkers of Thrombosis in ST-Segment Elevation Myocardial Infarction: A Substudy of the ATOLL Trial Comparing Enoxaparin Versus Unfractionated Heparin. Am J Cardiovasc Drugs. 2018 Dec;18(6):503-511. doi: 10.1007/s40256-018-0294-z. PMID 30144017